CLINICAL TRIAL: NCT04255667
Title: Outcome of Eyelid Crush for Intraoperative Hemostasis of Eyelid Margin Surgery
Brief Title: Eyelid Crush for Marginal Eyelid Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Tarek Roshdy mohamed Mahgoub ELhamaky, lecturer ophthalmology, Benha University
Other Study IDs: hamaky4
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Eyelid Diseases
Keywords: eyelid margin; hemostasis
MeSH Terms: conditions — Eyelid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Eyelid surgery involving eyelid margin is done after eyelid margin crushing with hemostat at start of surgery
  Interventions: Procedure: Eyelid margin crush
- Control group: Eyelid surgery involving eyelid margin is done after eyelid margin crushing without hemostat
  Interventions: Procedure: Eyelid margin crush

INTERVENTIONS:
Procedure: Eyelid margin crush — after marking eyelid , hemostat is used for eyelid margin incision crush . Then eyelid surgery is done

SUMMARY:
Surgery involves eyelid margin asscocited with intraoperative bleeding. Proper intra-operative homeostasis is essential for good intraoperative procedure and postoperative results.

DETAILED DESCRIPTION:
baseline and postoperative full ophthalmic examination was done.Procedure include all surgeries involving eyelid margin

ELIGIBILITY:
Inclusion Criteria:

* All surgeries involving eyelid margin

Exclusion Criteria:

* bleeding tendency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patient with marginal eyelid diseases surgeries will undergo surgeries
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
amount of intraoperative bleeding | intraoperative
  bleeding is recorded by photography

SECONDARY OUTCOMES:
time of operation | intraoperative
  time of surgery is recorded by stopwatch

CONTACTS AND LOCATIONS:
Overall Officials: TAREK R ELHAMAKY, MD, Principal Investigator — Benha university faculty of medicine
Locations (1):
- INMC, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No